CLINICAL TRIAL: NCT05639153
Title: An Open, Phase I, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of DR30303 in Patients With Advanced Solid Tumors
Brief Title: A Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of DR30303 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Doer Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR30303-101
Record Dates: First submitted 2022-11-08; First posted 2022-12-06 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Malignant Neoplasm of Digestive System
Keywords: Malignant neoplasm of digestive system
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DR30303 (Experimental): DR30303 injection treatment. This phase 1 trial will include two stages, a dose escalation stage and an expansion stage.
  Interventions: Drug: DR30303

INTERVENTIONS:
Drug: DR30303 — DR30303 dose level of escalation IV every 3 weeks (Q3W) Day 1, as well as dose expansion with recommended dose level from dose escalation.

SUMMARY:
This study is an open-label Phase 1, First in Human trial of DR30303, a recombinant humanized monoclonal antibody that targets Claudin18.2 (CLDN18.2). It is composed of humanized variable domain of heavy chain of antibody (VHH) fused with engineered immunoglobulin gamma-1(IgG1) Fc. It is being testing against advanced and/or metastatic solid tumors.

DETAILED DESCRIPTION:
This study is an open, phase I study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of DR30303 in patients with advanced solid tumors. The study is composed of two parts: part 1 is Dose escalation stage and part 2 is Dose expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed of this study and voluntarily sign informed consent form (ICF).
2. Aged 18 to 75 years, gender is not limited.
3. Part 1: Dose escalation stage - the subject have histologically or cytologically confirmed locally advanced or metastatic malignant solid tumors who have failed or are intolerant to prior systemic therapy.
4. Part 2: Dose expansion stage- CLDN18.2 positive confirmed by central laboratory locally advanced unresectable or metastatic gastric cancer (GC)/gastroesophageal junction (GEJ ) or Pancreatic cancer those who had failed or were intolerant to at least 1 line of systemic therapy.
5. The Eastern Cooperative Oncology Group (ECOG) score is 0 to 1.
6. Expected survival ≥ 3 months.
7. Adequate organ function.
8. Referring to the RECIST 1.1 standard, there is at least one measurable lesion.

Exclusion Criteria:

1. Radical radiotherapy was performed within 12 weeks before the first dose of study drug.
2. Subjects who have received other systemic anti-tumor therapy within 4 weeks before the first dose of study drug.
3. Subjects who received or are scheduled to receive live attenuated vaccine within 4 weeks.
4. Received systemic steroids equivalent to >10mg/d prednisone within 2 weeks before the first dose of study drug, except inhaled steroids.
5. Subjects who have undergone or are expected to undergo major surgery, or have severe unhealed wounds, etc. prior to the first dose of study drug.
6. Ever received any treatments targeting Claudin18.2.
7. Subject who have a history of allergy to any component in the DR30303.
8. Subject with uncontrolled intracranial metastases.
9. Uncontrollable pleural effusion, pericardial effusion and ascites effusion existed before enrollment.
10. hepatitis B virus (HBV), hepatitis C virus (HCV), HIV or syphilis infection.
11. Diseases or associated risks that are judged by the investigator to be inappropriate for enrollment, such as poorly controlled diabetes,etc.
12. Subjects with interstitial lung disease requiring treatment such as oral or intravenous corticosteroids.
13. Subjects with previous or concomitant malignancies, with the following exceptions: non- melanoma skin carcinoma in situ, superficial bladder cancer, etc.
14. Clinically significant cardiovascular and cerebrovascular diseases within 6 months before the first dose of study drug, such as New York Heart Association (NYHA) class III or IV congestive heart failure, etc.
15. Female patients who are breastfeeding.
16. The investigator assesses that the subject is unable or unwilling to comply with the requirements of the research protocol.
17. Participated in other clinical studies within the past 4 Weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1：Incidence of dose limiting toxicities (DLTs) | up to 21 days following first dose
Part 1：Number, severity and duration of treatment-emergent adverse events (TEAEs) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 | up to 28 days following last dose
Part 1：Maximum Tolerated Dose (MTD) and/or Biological effective dose (BED) based on safety, tolerability, PK profile and preliminary efficacy data | from date of last dose until the date of will receive DR30303 for 1 year or last documented progression，whichever occurs first
Part 2: Recommended Phase 2 Dose (RP2D) based on safety, tolerability, PK profile, and preliminary efficacy data | from date of first dose start until the date of first documented progression，or the date of death from any cause, or the date of will receive DR30303 for 1 year whichever came first
Part 2: Number, severity and duration of treatment-emergent adverse events (TEAEs) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 | up to 28 days following last dose

SECONDARY OUTCOMES:
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | from date of first dose start until the date of first documented progression，or the date of death from any cause, or the date of will receive DR30303 for 1 year whichever came first
  These measure are defined as the proportion of subjects with complete response (CR) or partial response (PR)
Disease control rate (DCR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | from date of first dose start until the date of first documented progression，or the date of death from any cause, or the date of will receive DR30303 for 1 year whichever came first
  These measure are defined as the proportion of subjects with CR, PR and stable disease (SD)
Duration of response (DOR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | from date of first dose start until the date of first documented progression，or the date of death from any cause, or the date of will receive DR30303 for 1 year whichever came first
  These measure are defined as the duration from the first occurrence of confirmed CR or PR until the date of disease progression or death (from any cause)
Clinical Benefit Rate | from date of first dose start until the date of first documented progression，or the date of death from any cause, or the date of will receive DR30303 for 1 year whichever came first
  Defined as Proportion of subjects with CR, PR and duration of SD ≥ 12 weeks
Duration of disease control (DDC) per RECIST v1.1 | from date of first dose start until the date of first documented progression，or the date of death from any cause, or the date of will receive DR30303 for 1 year whichever came first
  For subjects with CR, PR, or SD, duration was calculated from the first assessment as CR, PR, or SD until the date of disease progression or death (from any cause)
Progression free survival (PFS) per RECIST v1.1 | from date of first dose start until the date of first documented progression，or the date of death from any cause, or the date of will receive DR30303 for 1 year whichever came first
  These measure are defined as time from start of treatment to tumor progression or death from any cause
6-month and 12-month survival rates | from date of first dose start until the date of first documented progression , 6 months，12 months whichever came first
Overall survival (OS) per RECIST v1.1 | from date of first dose start until the date of first documented progression or death from any cause，or the date of will receive DR30303 for 1 year whichever came first
  These measure are defined as time from start of treatment to death from any cause
Pharmacokinetic (PK) of DR30303: Maximum serum concentration (Cmax) | up to 28 days following last dose
PK of DR30303: Area Under the concentration-time Curve from time zero to the last quantifiable concentration (AUC0-last) | up to 28 days following last dose
PK of DR30303: Area Under the concentration-time Curve from time zero to infinity (AUC0-inf) | up to 28 days following last dose
PK of DR30303: Time of the maximum concentration (tmax) | up to 28 days following last dose
PK of DR30303: Terminal elimination half-life (t1/2) | up to 28 days following last dose
Immunogenicity by measurement of Incidence of anti-drug antibodies (ADA) | up to 28 days following last dose

CONTACTS AND LOCATIONS:
Overall Officials: Hongming Pan, MD,PhD, Principal Investigator — Sir Run Run Shaw Hospital; Yanshan Huang, PhD, Study Chair — Zhejiang Doer Biologics Co., Ltd.; Junfang Xu, MD, Study Director — Huadong Medicine Co., Ltd.
Locations (1):
- Sir Run Run Shaw Hospital，Zhejiang University School of Medicine, Hanzhou, Zhejiang, China